CLINICAL TRIAL: NCT01383928
Title: An Open-Label, Dose-Escalation, Phase 1/2 Study of the Oral Formulation of IXAZOMIB (MLN9708), Administered Twice-weekly in Combination With Lenalidomide and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Requiring Systemic Treatment
Brief Title: Study of Oral IXAZOMIB in Combination With Lenalidomide and Dexamethasone in Participants With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16008; U1111-1168-1172 (Registry Identifier: WHO (UTN))
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Ixazomib 3 mg or 3.7 mg (Experimental): Ixazomib (MLN9708), orally, twice-weekly in combination with lenalidomide orally and dexamethasone orally as prescribed, in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 1. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly in 21-day treatment cycles as maintenance therapy until progressive disease or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Phase 2: Ixazomib 3 mg (Experimental): Ixazomib (MLN9708), orally, twice-weekly in combination with lenalidomide orally and dexamethasone orally as prescribed, in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 2. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly in 21-day treatment cycles as maintenance therapy until progressive disease or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
Drug: Lenalidomide — Lenalidomide capsules
Drug: Dexamethasone — Dexamethasone Tablets

SUMMARY:
The purpose of this study is to determine the safety, tolerability, maximum tolerated dose (MTD), and recommended phase 2 dose (RP2D) in phase 1 and to determine the combined response rate of clinical response CR and very good partial response (VGPR) in phase 2 of oral (PO) ixazomib administered twice-weekly in combination with lenalidomide and low-dose dexamethasone in a 21-day cycle in participants with newly diagnosed multiple myeloma (NDDM).

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib. Ixazomib was tested to slow disease progression and improve overall survival in participants who have newly diagnosed multiple myeloma (NDMM). This study looked at the safety, tolerability and response in participants when administered in combination with lenalidomide and low-dose dexamethasone.

The study enrolled 64 patients. Participants were assigned to one of the 3 treatment groups:

* Phase 1 Ixazomib 3 mg
* Phase 1 Ixazomib 3.7 mg
* Phase 2 Ixazomib 3 mg

All participants were administered with Ixazomib capsules, orally, twice-weekly on Days 1, 4, 8, and 11 along with lenalidomide capsules, orally, once daily on Days 1-14 and dexamethasone, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 1. Participants with stable or responding disease continued receiving ixazomib capsules, orally, twice weekly on Days 1, 4, 8, and 11 in 21-day treatment cycles as maintenance therapy until progressive disease or unacceptable toxicity.

This multi-center trial conducted in the United States. The overall time to participate in this study was 2037 days. Participants will make multiple visits to the clinic, and a final visit after 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Symptomatic multiple myeloma or asymptomatic myeloma with myeloma-related organ damage diagnosed according to standard criteria
* Measurable disease as specified in study protocol
* Hematologic, liver, and renal function as specified in the study protocol.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or agree to abstain from heterosexual intercourse; must also adhere to the guidelines of the lenalidomide pregnancy prevention program
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse AND must adhere to the guidelines of the lenalidomide pregnancy prevention program
* Must be able to take concurrent aspirin 325 mg daily
* Voluntary written consent

Exclusion Criteria

* Peripheral neuropathy that is greater or equal to Grade 2
* Female patients who are lactating or pregnant
* Major surgery or radiotherapy within 14 days before the first dose of study drug
* Uncontrolled infection requiring systematic antibiotics within 14 days before the first dose of study drug
* Diarrhea (> Grade 1)
* Prior systemic therapy for multiple myeloma, including investigational drugs (prior treatment with corticosteroids or localized radiation therapy dose not disqualify the patient)
* Systemic treatment with strong inhibitors of CYP1A2, strong inhibitors of CYP3A, or strong CYP3A inducers, or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study treatment
* Central nervous system involvement
* Diagnosis of smoldering multiple myeloma, Waldenstrom's macroglobulinemia, POEMS syndrome, plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome
* Evidence of current uncontrolled cardiovascular conditions
* Prior or concurrent deep vein thrombosis or pulmonary embolism
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol
* Known allergy to any of the study medications
* Known gastrointestinal condition or procedure that could interfere with swallowing or the oral absorption, or tolerance of IXAZOMIB
* Diagnosed or treated for another malignancy within 2 years before the first dose or previously diagnosed with another malignancy and have any evidence of residual disease with the exception of nonmelanoma skin cancer or any completely resected carcinoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2014-10-13 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (20):
- United States (20):
  - UCSF Medical Center, Berkeley, California
  - City of Hope National Medical Center, Duarte, California
  - Stanford University, Stanford, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Associates of Oncology/Hematology PC, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, Lansing, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Mercy St Anne Hospital, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - SCRI Tennessee Oncology Nashville, Nashville, Tennessee
  - Baylor Sammons Cancer Center, Dallas, Texas
  - Virginia Cancer Care Specialist, Fairfax, Virginia
  - Virginia Cancer Specialists PC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 15 investigative sites in the United States from 31 October 2011 to 27 November 2017 when the sponsor closed the study.
Pre-assignment Details: Participants with newly diagnosed multiple myeloma were enrolled in 1 of the 2 dose escalation treatment arms in Phase 1: ixazomib 3 mg and 3.7 mg induction followed by maintenance. Phase 2 consisted of ixazomib 3 mg during induction followed by maintenance.
Groups:
- Phase 1: Ixazomib 3 mg: Ixazomib 3 mg, capsules, orally, twice-weekly on Days 1, 4, 8, and 11, lenalidomide 25 mg, capsules, orally, once daily on Days 1-14, dexamethasone 20 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 in Cycle 1-8 and dexamethasone 10 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 in Cycle 9-16 in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 1. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly on Days 1, 4, 8, and 11 in 21-day treatment cycles as maintenance therapy at the dose tolerated at the end of induction until progressive disease or unacceptable toxicity. The maximum number of cycles received was 83 cycles (approximately up to 2037 days).
- Phase 1: Ixazomib 3.7 mg: Ixazomib (MLN9708) 3.7 mg, capsules, orally, twice-weekly on Days 1, 4, 8, and 11, lenalidomide 25 mg, capsules, orally, once daily on Days 1-14, dexamethasone 20 mg, capsules, orally, once daily on days 1, 2, 4, 5, 8, 9, 11, and 12 in Cycle 1-8 and dexamethasone 10 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 in Cycle 9-16 in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 1. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly on Days 1, 4, 8, and 11 in 21-day treatment cycles as maintenance therapy at the dose tolerated at the end of induction until progressive disease or unacceptable toxicity. The maximum number of cycles received in this cohort was 25 cycles (approximately 585 days).
- Phase 2: Ixazomib 3 mg: Ixazomib 3 mg (MLN9708), capsules, orally, twice-weekly on Days 1, 4, 8, and 11, lenalidomide 25 mg capsules, orally, once daily on Days 1-14, dexamethasone 20 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11 and 12 in Cycle 1-8 and dexamethasone 10 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11 and 12 in Cycle 9-16 in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 2. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly on Days 1, 4, 8, and 11 in 21-day treatment cycles as maintenance therapy at the dose tolerated at the end of induction until progressive disease or unacceptable toxicity. The maximum number of cycles received in this cohort was 74 cycles (approximately 1875 days).
Period: Overall Study
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg | Phase 2: Ixazomib 3 mg
Started | 7 | 7 | 50
Completed (Completed=participants who completed 16 cycles per protocol and entered Maintenance phase.) | 2 | 0 | 10
Not Completed | 5 | 7 | 40
Not completed — Initiation of ASCT | 2 | 1 | 18
Not completed — Adverse Event | 1 | 2 | 8
Not completed — Other | 1 | 3 | 4
Not completed — Progressive Disease | 1 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Unsatisfactory Therapeutic Response | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg | Phase 2: Ixazomib 3 mg | Total
Number analyzed (Participants) | 7 | 7 | 50 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (12.04) | 61.1 (6.20) | 61.5 (10.03) | 61.8 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 19 | 24
  Male | 5 | 4 | 31 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 7 | 48 | 62
  Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 7 | 42 | 54
  Black or African American | 1 | 0 | 7 | 8
  Other | 1 | 0 | 0 | 1
  Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 50 | 64
Height [Mean (Standard Deviation); unit: cm] — Population: For this baseline measure, number of participants evaluable were 7, 6 and 49 for each arm, respectively.
  cm
    number analyzed (Participants) | 7 | 6 | 49 | 62
    (all) | 171.1 (13.09) | 170.9 (7.10) | 171.2 (9.30) | 171.1 (9.43)
Weight [Mean (Standard Deviation); unit: kg] | 94.29 (17.083) | 82.56 (19.295) | 81.22 (16.701) | 82.80 (17.228)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: For this baseline measure, number of participants evaluable were 7, 6 and 49 for each arm, respectively.
  m^2
    number analyzed (Participants) | 7 | 6 | 49 | 62
    (all) | 2.109 (0.2192) | 1.960 (0.2657) | 1.958 (0.2373) | 1.975 (0.2390)
Type of Myeloma [Count of Participants; unit: Participants] — Types of Myeloma was described on the basis of antibodies produced by cancerous plasma cells.
  Participants
    IgG Kappa | 2 | 3 | 24 | 29
    IgG Lambda | 1 | 1 | 7 | 9
    IgA Kappa | 1 | 1 | 10 | 12
    IgA Lambda | 1 | 0 | 3 | 4
    Biclonal | 0 | 1 | 1 | 2
    Lambda Free Light Chains | 1 | 0 | 3 | 4
    Kappa Free Light Chains | 1 | 1 | 1 | 3
    Unknown | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to assess how the disease affects the daily living abilities of the participant. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead.
  Participants
    0 | 3 | 5 | 27 | 35
    1 | 4 | 1 | 21 | 26
    2 | 0 | 1 | 2 | 3
Serum Creatinine Category [Count of Participants; unit: Participants]
  Less than or equal to (<=) 2 mg/dL | 7 | 7 | 50 | 64
  Greater than (>) 2 mg/dL | 0 | 0 | 0 | 0
Creatinine Clearance Category [Count of Participants; unit: Participants]
  30 - 60 mL/min | 2 | 2 | 8 | 12
  >60 mL/min | 5 | 5 | 42 | 52
Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] — Corrected calcium was calculated using the following formula: serum calcium (mg/dL)+0.98*[4-serum albumin (gram per deciliter [g/dL])]
  mg/dL | 9.83 (0.275) | 9.79 (0.561) | 10.01 (0.617) | 9.96 (0.583)
Hemoglobin [Mean (Standard Deviation); unit: gram per liter (g/L)] | 103.4 (21.59) | 112.0 (16.42) | 108.9 (14.36) | 108.6 (15.32)
Participants with Lytic Bone Lesions Present [Count of Participants; unit: Participants]
  Present | 5 | 3 | 37 | 45
  Not Present | 1 | 2 | 7 | 10
  Indeterminate | 0 | 0 | 1 | 1
  Missing | 1 | 2 | 5 | 8
Participants with Extramedullary Plasmacytomas [Count of Participants; unit: Participants] — Population: Participants who performed magnetic resonance imaging (MRI)/computed tomography (CT) scan were eligible for this baseline measure.
  Participants
    Plasmacytomas Present | 1 | 1 | 18 | 20
    Plasmacytomas Not Present | 2 | 2 | 4 | 8
    Not Reported | 4 | 4 | 28 | 36

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)
Description: MTD was highest dose of ixazomib given with combination drugs, at which <=1 of 6 participants experienced dose-limiting toxicity (DLT) during Cycle 1 of Phase 1. DLT defined as any of following considered possibly related to therapy: Grade 4 neutropenia (absolute neutrophil count [ANC] <500 cell per cubic millimeter [cells/mm^3]) for >7 days; Grade 3 neutropenia with fever or infection; Grade 4 thrombocytopenia for >7 days; Grade 3 thrombocytopenia with clinically significant bleeding; platelet count <10,000/mm^3; Grade 2 peripheral neuropathy with pain or >=Grade 3 peripheral neuropathy; >=Grade 3 nausea/emesis, diarrhea controlled by supportive therapy; any >=Grade 3 nonhematologic toxicity except Grade 3 arthralgia/myalgia; or <1 week Grade 3 fatigue; delay in initiation of the subsequent therapy cycle by >14 days; <=80% lenalidomide doses administered due to other >=Grade 2 combination study drug-related nonhematologic toxicities requiring therapy discontinuation.
Time Frame: Cycle 1 (21 days)
Population: DLT-evaluable population included all participants who received all Cycle 1 doses of MLN9708 and completed Cycle 1 procedures, or experienced a DLT in Cycle 1 in Phase 1.
Measure: Number; unit: mg
Groups:
- Phase 1: All Participants: Ixazomib 3 mg or 3.7 mg, capsules, orally, twice-weekly on Days 1, 4, 8, and 11, lenalidomide 25 mg, capsules, orally, once daily on Days 1-14, dexamethasone 20 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 in Cycle 1-8 and dexamethasone 10 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 in Cycle 9-16 in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 1. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly on Days 1, 4, 8, and 11 in 21-day treatment cycles as maintenance therapy at the dose tolerated at the end of induction until progressive disease or unacceptable toxicity. The maximum number of cycles received was 83 cycles (approximately up to 2037 days).
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 14
mg | 3.7

2. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D)
Description: The RP2D of ixazomib was determined after the evaluation of the available data from the phase 1 portion of the trial which included, but was not limited to analyses of efficacy results, toxicity characterization, all grades peripheral neuropathy, and treatment discontinuation. The maximum number of cycles received was 83 cycles (approximately up to 2037 days).
Time Frame: Cycle 1 (21 days)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: mg
Arm/Group | Phase 1: All Participants
Number analyzed (Participants) | 14
mg | 3

3. Primary Outcome: Phase 1: Percentage of Participants Experiencing 1 or More Treatment-Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 30 days after last dose of study drug (Up to Cycle 83 - approximately 2067 days)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 7 | 7
percentage of participants
  Adverse Event | 100 | 100
  Serious Adverse Event | 71 | 29

4. Primary Outcome: Phase 1: Number of Participants With Markedly Abnormal Laboratory Values Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Laboratory tests included chemistry, hematology and urinalysis. Abnormal laboratory value was assessed as an AE if the value lead to discontinuation or delay in treatment, dose modification, therapeutic intervention, or was considered by the investigator to be a clinically significant change from baseline. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 30 days after last dose of study drug (Up to Cycle 83 - approximately 2067 days)
Population: Safety population included all participants who received at least 1 dose of any study drug and reported baseline and at least 1 post-baseline value.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 7 | 7
Participants
  Alanine aminotransferase increased | 0 | 3
  Aspartate aminotransferase increased | 0 | 2
  Blood creatinine increased | 2 | 0
  Shift to the left | 0 | 1
  Platelet count decreased | 1 | 0
  Blood bicarbonate decreased | 1 | 0
  Anaemia | 1 | 0
  Neutropenia | 1 | 0
  Thrombocytopenia | 1 | 1
  Eosinophilia | 0 | 1
  Hypokalaemia | 1 | 0
  Hyperkalaemia | 1 | 0
  Hyperglycaemia | 4 | 0
  Hyponatraemia | 0 | 1
  Hypomagnesaemia | 0 | 2
  Hyperchloraemia | 1 | 0
  Iron deficiency anaemia | 1 | 0

5. Primary Outcome: Phase 1: Number of Participants With Treatment-Emergent Adverse Events (TEAE) Related to Neurotoxicity
Description: TEAE related to neurotoxicity grading based on common terminology criteria for adverse events (CTACE) version 4.03 are reported. Grade 1= mild; Grade 2= moderate; within normal limits, Grade 3= severe or medically significant but not immediately life-threatening; Grade 4= life-threatening consequences; urgent intervention indicated; Grade 5= death. Only TEAEs related to neurotoxicity with values are reported.
Time Frame: Baseline up to 30 days after last dose of study drug (Up to Cycle 83 - approximately 2067 days)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 7 | 7
Participants
  Neuropathy Peripheral (Grade 1) | 0 | 1
  Neuropathy Peripheral (Grade 2) | 2 | 1
  Neuropathy Peripheral (Grade 3) | 0 | 1
  Peripheral Sensory Neuropathy (Grade 1) | 2 | 1
  Peripheral Sensory Neuropathy (Grade 2) | 0 | 1
  Peripheral Sensory Neuropathy (Grade 3) | 1 | 0
  Peripheral Motor Neuropathy (Grade 1) | 1 | 0

6. Primary Outcome: Phase 1: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature, blood pressure and heart rate.
Time Frame: Baseline up to 30 days after last dose of study drug (Up to Cycle 83 - approximately 2067 days)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 7 | 7
Participants
  Pyrexia | 1 | 3
  Bradycardia | 1 | 0
  Orthostatic hypotension | 0 | 1
  Hypotension | 1 | 1

7. Primary Outcome: Phase 2: Percentage of Participants With Complete Response (CR) + Very Good Partial Response (VGPR)
Description: CR as per International Myeloma Working Group (IMWG) uniform criteria is defined as negative immunofixation on the serum and urine and disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow. VGPR as per IMWG criteria is defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours. VGPR was applicable only to participants who had measurable disease defined by at least 1 of the following 3 measurements: Serum M-protein greater than or equal to (>=)1 g/dL; Urine M-protein >=200 mg/24 hours; Serum FLC assay level >=10 mg/dL, provided serum FLC ratio was abnormal.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: Response-evaluable population included all participants who received at least 1 dose of study drug, had measurable disease at baseline, and at least 1 post-baseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 65 [50.4 to 78.3]

8. Primary Outcome: Phase 2: Percentage of Participants With Grade 3 or Higher Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. As per Common Terminology Criteria for Adverse Events v4.0 (CTCAE), Grade 3 = AE with severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4 = AE with life-threatening consequences; urgent intervention indicated and Grade 5 = Death related to AE.
Time Frame: Baseline up to 30 days after the last dose of study drug (approximately 1905 days)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 50
percentage of participants | 74

9. Primary Outcome: Phase 2: Percentage of Participants Experiencing Serious Adverse Events
Description: A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: Baseline up to 30 days after the last dose of study drug (approximately 1905 days)
Population: Safety population included all participants who received at least one dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 50
percentage of participants | 46

10. Primary Outcome: Phase 2: Percentage of Participants With Treatment-Emergent Adverse Events Resulting in Study Drug Discontinuation
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 30 days after the last dose of study drug (approximately 1905 days)
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 50
percentage of participants | 14

11. Secondary Outcome: Phase 1: Cmax: Maximum Plasma Concentration for Ixazomib
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of ixazomib, obtained directly from the plasma concentration-time curve.
Time Frame: Cycle 1, Days 1 and 11
Population: Pharmacokinetic (PK) analysis population included all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters where Days 1 and 11 assessments were available.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 7 | 7
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 6 | 7
  Day 1 | 33.515 (22.9634) | 46.946 (26.6436)
  Day 11: number analyzed (Participants) | 7 | 6
  Day 11 | 58.674 (19.9559) | 51.832 (23.5112)

12. Secondary Outcome: Phase 1: AUC(0-72): Area Under the Plasma Concentration-Time Curve From Time 0 to 72 Hours Postdose for Ixazomib
Description: AUC(0-72) is a measure of the area under the plasma concentration time-curve from time zero to 72 hours post-dose for ixazomib.
Time Frame: Cycle 1, Days 1 and 11
Population: PK analysis population included all participants, who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters where Days 1 and 11 assessments were available.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 7 | 7
hour*nanogram per milliliter (hr*ng/mL)
  Day 1: number analyzed (Participants) | 5 | 6
  Day 1 | 315.450 (75.0886) | 284.576 (47.8233)
  Day 11: number analyzed (Participants) | 7 | 6
  Day 11 | 1105.44 (457.5939) | 1023.52 (284.3709)

13. Secondary Outcome: Phase 1: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Description: Tmax: Time to reach the first maximum plasma concentration (Cmax), equal to time (hours) to Cmax of ixazomib after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Cycle 1, Days 1 and 11
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 7 | 7
hours
  Day 1: number analyzed (Participants) | 6 | 7
  Day 1 | 1.035 [0.53 to 1.60] | 1.000 [0.50 to 1.47]
  Day 11: number analyzed (Participants) | 7 | 6
  Day 11 | 1.030 [0.50 to 4.00] | 0.984 [0.50 to 2.08]

14. Secondary Outcome: Phase 1: Rac: Accumulation Ratio of Ixazomib
Description: The accumulation ratio (Rac) was estimated as the ratio of AUC (0-72) on Day 11 to the AUC (0-72) on Day 1. AUC (0-72) is the area under the plasma concentration-time curve from time zero to 72 hours post-dose for ixazomib.
Time Frame: Cycle 1, Days 1 and 11
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg
Number analyzed (Participants) | 5 | 5
ratio | 3.785 (1.4653) | 3.967 (0.7546)

15. Secondary Outcome: Phase 1: Percentage of Participants With Best Overall Response
Description: CR as per International Myeloma Working Group (IMWG) uniform criteria is defined as negative immunofixation on the serum and urine and disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow. Partial response(PR):>=50% reduction of serum M-protein,urinary M-protein by >=90%/to <200 mg/24 hr reduction.Near CR(nCR):positive immunofixation of serum/urine;soft tissue plasmacytomas disappearance;<=5% plasma cells in bone marrow. VGPR as per IMWG criteria is defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours. VGPR was applicable only to participants who had measurable disease defined by at least 1 of the following 3 measurements: Serum M-protein greater than or equal to (>=)1 g/dL; Urine M-protein >=200 mg/24 hours; Serum FLC assay level >=10 mg/dL, provided serum FLC ratio was abnormal.
Time Frame: Baseline until end of study treatment (Up to treatment Cycle 83 - approximately 2037 days)
Population: Response-evaluable population included all participants who received at least 1 dose of ixazomib, had measurable disease at baseline, and at least 1 post-baseline disease assessment. Results were summarized together for all Phase 1 participants, as per planned analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Ixazomib 3 mg
Number analyzed (Participants) | 13
percentage of participants | 92 [64 to 99.8]

16. Secondary Outcome: Phase 2: Percentage of Participants With Overall Response (CR+VGPR+PR)
Description: Overall response is defined as CR, VGPR or PR based on IMWG Response Criteria for malignant lymphoma. CR: disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. VGPR: serum, urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein+urine M-protein level <100 mg/24h. Partial response (PR) is a minimum of 50% decrease in sum of the product of the diameters of up to 6 of the largest dominant nodes or nodal masses and no increase in the size of other nodes.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: Response-evaluable population included all participants who received at least 1 dose of ixazomib, had measurable disease at baseline, and at least 1 post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 94 [83.1 to 98.7]

17. Secondary Outcome: Phase 2: Percentage of Participants With Complete Response (CR) and Very Good Partial Response (VGPR) After Cycles 4, 8, and 16
Description: CR as per IMWG criteria is defined as negative immunofixation on the serum and urine and disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow. VGPR as per IMWG criteria is defined as serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours. VGPR were applicable only to participants who had measurable disease defined by at least 1 of the following 3 measurements: Serum M-protein; Urine M-protein; Serum FLC assay.
Time Frame: Cycles 4, 8, and 16
Population: Response-evaluable population included all participants who received at least one 1 dose of ixazomib, had measurable disease at baseline, and at least one 1 post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants
  After 4 cycles | 49 [34.1 to 63.9]
  After 8 cycles | 64 [42.5 to 82.0]
  After 16 cycles | 92 [61.5 to 99.8]

18. Secondary Outcome: Phase 2: Percentage of Participants With Complete Response (CR)
Description: CR as per IMWG criteria is negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 29 [16.6 to 43.3]

19. Secondary Outcome: Phase 2: Percentage of Participants With Stringent Complete Response (sCR)
Description: sCR as per IMWG criteria is CR plus normal FLC ratio and absence of clonal cells in bone marrow. CR is negative immunofixation on serum and urine and disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 22 [11.8 to 36.6]

20. Secondary Outcome: Phase 2: Percentage of Participants With Very Good Partial Response (VGPR)
Description: VGPR as per IMWG criteria is serum and urine M-protein detectable by immunofixation but not on electrophoresis or >=90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 37 [23.4 to 51.7]

21. Secondary Outcome: Phase 2: Percentage of Participants With Near Complete Response (nCR)
Description: nCR as per IMWG criteria is positive immunofixation analysis of serum or urine as the only evidence of disease; appearance of any soft tissue plasmacytomas and <=5% plasma cells in bone marrow.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 10 [3.4 to 22.2]

22. Secondary Outcome: Phase 2: Percentage of Participants With Partial Response (PR)
Description: PR as per IMWG criteria is 50% reduction of serum M-protein and reduction in 24-hr urinary M-protein by 90% or to <200 mg per 24 hours.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 65 [50.4 to 78.3]

23. Secondary Outcome: Phase 2: Percentage of Participants With Minimal Response (MR)
Description: MR as per IMWG criteria is 25%-49% reduction in serum paraprotein and 50%-89% reduction in urine light chain excretion for 6 weeks.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
percentage of participants | 6 [1.3 to 16.9]

24. Secondary Outcome: Phase 2: Time to Response
Description: Time to first response is defined as the time from the date of first dose of study treatment to the date of the first documentation of a confirmed response (PR or better) in a participant who responded + 1 day. PR as per IMWG criteria is 50% reduction of serum M-protein and reduction in 24-h urinary M-protein by 90% or to <200 mg per 24 hours.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 46
months | 0.72 [0.7 to 4.5]

25. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was measured as the time from the date of first documentation of a confirmed response to the date of first documented PD. PD is defined as >=25% increase from lowest value in: serum/urine M-component; difference between involved, uninvolved FLC levels; bone marrow plasma cell percent; development of new bone lesions or soft tissue plasmacytomas development or increase in the size of existing bone lesions or soft tissue plasmacytomas; hypercalcaemia development.
Time Frame: Baseline until end of treatment (Up to treatment Cycle 74 - approximately 1875 days)
Population: Included a subset of response-evaluable population who achieved response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ixazomib 3 mg
Number analyzed (Participants) | 49
months | 29.0 [16.72 to NA] — Upper limit of 95% confidence interval was not estimable as majority of the participants were censored.

26. Secondary Outcome: Time to Disease Progression (TTP)
Description: Time to progression was defined as the time from the date of first dose of study treatment to the date of first documentation of PD + 1 day. Participants that did not experience PD will be censored at the last response assessment that is SD or better. PD: >=25% increase from lowest value in:serum/urine M-component; difference between involved, uninvolved FLC levels; bone marrow plasma cell percent; new bone lesions/soft tissue plasmacytomas development/existing bone lesions/soft tissue plasmacytomas size rise; hypercalcaemia development. SD: not meeting criteria for CR, VGPR, PR, or PD. Participants that received Autologous Stem Cell Transplantation (ASCT) or an alternate cancer therapy were also be censored at the last response assessment that is, SD or better prior to initiation of therapy. Participants without response assessment will be censored at the date of first dose. TTP was analyzed using standard survival analysis techniques based on Kaplan-Meier estimates.
Time Frame: Baseline up to a follow-up of 62.1 months
Population: modified-intent-to-treat (mITT) population included all participants who received at least one dose of any study drug in Phase 2 or who received at least 1 dose of any study drug and were treated at the phase 2 dose level during Phase 1.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ixazomib 3 mg: Ixazomib 3 mg (MLN9708), capsules, orally, twice-weekly on Days 1, 4, 8, and 11, lenalidomide 25 mg capsules, orally, once daily on Days 1-14, dexamethasone 20 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11 and 12 in Cycle 1-8 and dexamethasone 10 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11 and 12 in Cycle 9-16 in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 2. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly on Days 1, 4, 8, and 11 in 21-day treatment cycles as maintenance therapy at the dose tolerated at the end of induction until progressive disease or unacceptable toxicity. The maximum number of cycles received in this cohort was 83 cycles (approximately 2037 days).
Arm/Group | Ixazomib 3 mg
Number analyzed (Participants) | 57
months | 29.7 [17.41 to 66.0]

27. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of first dose of study treatment to the date of first documentation of progressive disease or to death due to any cause, whichever occurred first plus 1. PD: >=25% increase from lowest value in:serum/urine M-component; difference between involved,uninvolved FLC levels; bone marrow plasma cell percent; new bone lesions/soft tissue plasmacytomas development/existing bone lesions/soft tissue plasmacytomas size rise; hypercalcaemia development. SD: not meeting criteria for CR, VGPR, PR, or PD. Participants who received ASCT or an alternate anticancer therapy were censored at the last response assessment that was SD or better before initiation of therapy. Participants without a response assessment were censored at the date of first dose. PFS was analyzed using standard survival analysis techniques based on Kaplan-Meier estimates.
Time Frame: Baseline up to a follow-up of 62.1 months
Population: mITT population included all participants who received at least 1 dose of any study drug in Phase 2 or who received at least 1 dose of any study drug and were treated at the phase 2 dose level during Phase 1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 3 mg
Number analyzed (Participants) | 57
months | 29.7 [17.41 to 66.0]

28. Secondary Outcome: Kaplan-Meier Estimate of Percentage of Participants Achieving Survival at Year 1
Description: The Kaplan-Meier estimate reports the percentage of participants surviving at Year 1.
Time Frame: 1 year after the first dose of study treatment
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ixazomib 3 mg
Number analyzed (Participants) | 57
percentage of participants | 94 [84 to 98]

29. Secondary Outcome: Overall Survival
Description: Overall survival was measured as the time from the date of first dose of study treatment to the time of death plus 1 day. For participants who did not die, survival was censored at the date of last contact. Overall Survival was analyzed using standard survival analysis techniques based on Kaplan-Meier estimates.
Time Frame: Baseline up to a follow-up of 62.1 months
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixazomib 3 mg
Number analyzed (Participants) | 57
months | NA [60.19 to NA] — Median and upper limit of 95% confidence interval was not estimable as majority of the participants were censored.

ADVERSE EVENTS:
Time Frame: From first study drug administration up to 30 days after the last dose (Up to approximately 2067 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Phase 2: Ixazomib 3.0 mg: Ixazomib 3 mg (MLN9708), capsules, orally, twice-weekly on Days 1, 4, 8, and 11, lenalidomide 25 mg capsules, orally, once daily on Days 1-14, dexamethasone 20 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11 and 12 in Cycle 1-8 and dexamethasone 10 mg, capsules, orally, once daily on Days 1, 2, 4, 5, 8, 9, 11 and 12 in Cycle 9-16 in 21-day treatment cycles for up to 16 cycles in the absence of disease progression or unacceptable toxicity as induction therapy during Phase 2. Participants with stable or responding disease continued receiving ixazomib (MLN9708) orally, twice weekly on Days 1, 4, 8, and 11 in 21-day treatment cycles as maintenance therapy at the dose tolerated at the end of induction until progressive disease or unacceptable toxicity. The maximum number of cycles received in this cohort was 74 cycles (approximately 1875 days).
Arm/Group | Phase 1: Ixazomib 3 mg | Phase 1: Ixazomib 3.7 mg | Phase 2: Ixazomib 3.0 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 1/50
Serious Adverse Events (participants affected / at risk) | 5/7 | 2/7 | 23/50
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Ixazomib 3 mg (N=7) | Phase 1: Ixazomib 3.7 mg (N=7) | Phase 2: Ixazomib 3.0 mg (N=50)
Pneumonia (Infections and infestations) | 1 | 0 | 3
Lung infection (Infections and infestations) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 2
Skin infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Scrotal infection (Infections and infestations) | 1 | 0 | 0
Infective myositis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 — one treatment-emergent death occurred during study and is related to study drug.
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Ixazomib 3 mg (N=7) | Phase 1: Ixazomib 3.7 mg (N=7) | Phase 2: Ixazomib 3.0 mg (N=50)
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 23
Nausea (Gastrointestinal disorders) | 4 | 4 | 20
Constipation (Gastrointestinal disorders) | 2 | 3 | 20
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | 0
Palatal oedema (Gastrointestinal disorders) | 1 | 0 | 0
Tongue erythema (Gastrointestinal disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 4 | 4 | 22
Fatigue (General disorders) | 5 | 6 | 24
Asthenia (General disorders) | 2 | 0 | 9
Chills (General disorders) | 1 | 1 | 4
Pain (General disorders) | 1 | 0 | 5
Gait disturbance (General disorders) | 0 | 0 | 3
Localised oedema (General disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 2 | 20
Dizziness (Nervous system disorders) | 3 | 1 | 15
Tremor (Nervous system disorders) | 5 | 0 | 7
Hypoaesthesia (Nervous system disorders) | 2 | 2 | 7
Paraesthesia (Nervous system disorders) | 1 | 1 | 5
Ageusia (Nervous system disorders) | 1 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 2 | 1
Lethargy (Nervous system disorders) | 1 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 3
Presyncope (Nervous system disorders) | 0 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 1 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 7
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 4
Hyperchloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 6 | 17
Anxiety (Psychiatric disorders) | 2 | 1 | 13
Depression (Psychiatric disorders) | 0 | 1 | 4
Mood altered (Psychiatric disorders) | 0 | 0 | 4
Agitation (Psychiatric disorders) | 0 | 2 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 19
Sinusitis (Infections and infestations) | 1 | 1 | 8
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 7
Oral candidiasis (Infections and infestations) | 0 | 0 | 6
Oral herpes (Infections and infestations) | 0 | 0 | 4
Herpes zoster (Infections and infestations) | 0 | 1 | 2
Folliculitis (Infections and infestations) | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 15
Cataract (Eye disorders) | 0 | 0 | 5
Blood creatinine increased (Investigations) | 2 | 0 | 5
Weight decreased (Investigations) | 1 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 3
Weight increased (Investigations) | 0 | 0 | 4
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Shift to the left (Investigations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Flushing (Vascular disorders) | 2 | 2 | 3
Hot flush (Vascular disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 4
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 4
Bradycardia (Cardiac disorders) | 1 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2
Cushingoid (Endocrine disorders) | 1 | 0 | 2
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 6
Vomiting (Gastrointestinal disorders) | 3 | 0 | 13
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4
Enlarged uvula (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 0 | 8
Peripheral swelling (General disorders) | 1 | 0 | 9
Non-cardiac chest pain (General disorders) | 1 | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 4
Conjunctivitis (Infections and infestations) | 1 | 0 | 2
Skin infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 4
Platelet count decreased (Investigations) | 1 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 17
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 5 | 0 | 18
Headache (Nervous system disorders) | 6 | 0 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | 12
Balance disorder (Nervous system disorders) | 0 | 0 | 3
Syncope (Nervous system disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 6
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Hypotension (Vascular disorders) | 2 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.